CLINICAL TRIAL: NCT04642677
Title: Randomized phasE II Study for Efficacy of healThcare prOvider's REcommened Communication With Sympathy in Terminally Ill Cancer Patients Treated With Palliative Sedation
Brief Title: REcommened Communication With Sympathy in Terminally Ill Cancer Patients Treated With Palliative Sedation
Acronym: RESTORE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kwonoh Park, MD phD, Assistant professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESTORE
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Communication, Palliative Sedation
Keywords: Communication, Palliative sedation
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Prospective, Single institution, Open-label, Randomized, Phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients and caregivers were received palliative sedation with healthcare provider's recommended communication with sympathy and printed paper, "Regardless of the patient's outward consciousness, talk with the patient and express empathy. Hearing will be maintained until the end." three times a day (8, 14 and 20 o'clock).
  Interventions: Other: healthcare provider's recommended communication with sympathy and printed paper
- Group B (No Intervention): Patients and caregivers were received palliative sedation without intervention.

INTERVENTIONS:
Other: healthcare provider's recommended communication with sympathy and printed paper — Patients and caregivers were received healthcare provider's recommended communication with sympathy and printed paper, "Regardless of the patient's outward consciousness, talk with the patient and express empathy. Hearing will be maintained until the end." three times a day (8, 14 and 20 o'clock) during palliative sedation.
  Arms: Group A

SUMMARY:
* In terminally ill cancer patients, palliative sedation has been applied to intractable refractory symptoms such as pain, dyspnea, delirium, agitation.
* Palliative sedation is generally an adaptive strategies using midazolam, which is composed of intermittent bolus, limited continuous, or 24hr continuous infusion depending on the time of drug application.
* In the application of palliative sedation, caregiver's negative feelings such as anxiety or guilt for palliative sufficiency are one of the biggest challenges as the patient's consciousness is reduced, and they feels disconnected from the patient.
* In general, hearing is known to persist until the very last moment of the end of life, regardless of consciousness. In addition, maintaining communication with patients and caregivers is the most important part of the hospice.
* This study evaluate the efficacy of healthcare provider's recommended communication with sympathy, "Regardless of the patient's outward consciousness, talk with the patient and express empathy. Hearing will be maintained until the end."

ELIGIBILITY:
Inclusion Criteria:

* Patients who are expected to die within a few weeks due to disease progression without additional anti-tumor treatment plans.
* Patients who are the target of palliative sedation because intractable symptom such as pain, dyspnea, delirium, or agitation persist as even after the conservative treatment.
* Patients who have agreed to palliative sedation.

Exclusion Criteria:

* Patients treated with a palliative sedation methods using bolus application or other drugs (lorazepam, etc.) rather than continuous midazolam were excluded.
* In case of the guardian is unable to stay with the patient for more than 6 hours per day, the patients were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate of palliative sedation irrespective of physician | From date of enrollment until death or discharge/transfer, assess up to 2 years
  Rate of cases (caregiver's refuse or others) among all causes (death, multi-organ failure, failure of sedation level, palliative sedation related adverse events, caregiver's refuse, or others) as discontinuation causes of palliative sedation
Complete response rate of palliative sedation | From date of enrollment until death or discharge/transfer, assess up to 2 years
  Rate of cases (death or multiogran failure) among all causes (death, multi-organ failure, failure of sedation level, palliative sedation related adverse events, caregiver's refuse, or others) as discontinuation causes of palliative sedation

SECONDARY OUTCOMES:
Satisfaction of caregiver | 2th to 7th day after enrollment
  How is your satisfaction with the IV access so far?" (rated as "much comfort", "a little comfort", "no change", "a little discomfort", or "much discomfort")
Anxiety of caregiver | 2th to 7th day after enrollment
  GAD-7 (General Anxiety Disorder-7)
Palliative sedation related Adverse events | From date of enrollment until death or discharge/transfer, assess up to 2 years
  Adverse events related with palliative sedation using CTCAE 4.3

CONTACTS AND LOCATIONS:
Overall Officials: Kwonoh Park, MD, phD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Maltoni M, Scarpi E, Nanni O. Palliative sedation in end-of-life care. Curr Opin Oncol. 2013 Jul;25(4):360-7. doi: 10.1097/CCO.0b013e3283622c47. PMID 23666472
- [Result] Eun Y, Hong IW, Bruera E, Kang JH. Qualitative Study on the Perceptions of Terminally Ill Cancer Patients and Their Family Members Regarding End-of-Life Experiences Focusing on Palliative Sedation. J Pain Symptom Manage. 2017 Jun;53(6):1010-1016. doi: 10.1016/j.jpainsymman.2016.12.353. Epub 2017 Feb 10. PMID 28192224
- [Result] Kang JH, Shin SH, Bruera E. Comprehensive approaches to managing delirium in patients with advanced cancer. Cancer Treat Rev. 2013 Feb;39(1):105-12. doi: 10.1016/j.ctrv.2012.08.001. Epub 2012 Sep 6. PMID 22959227
- [Result] Maltoni M, Scarpi E, Rosati M, Derni S, Fabbri L, Martini F, Amadori D, Nanni O. Palliative sedation in end-of-life care and survival: a systematic review. J Clin Oncol. 2012 Apr 20;30(12):1378-83. doi: 10.1200/JCO.2011.37.3795. Epub 2012 Mar 12. PMID 22412129
- [Result] Papavasiliou EE, Payne S, Brearley S; EUROIMPACT. Current debates on end-of-life sedation: an international expert elicitation study. Support Care Cancer. 2014 Aug;22(8):2141-9. doi: 10.1007/s00520-014-2200-9. Epub 2014 Mar 20. PMID 24647491